CLINICAL TRIAL: NCT02976948
Title: Evaluation of a New Sequencing Strategy in Autoinflammatory Diseases Diagnostic Value and Therapeutic Orientation
Brief Title: Evaluation of a New Sequencing Strategy in Autoinflammatory Siseases (BIOSAID)
Acronym: BIOSAID
Status: Terminated | Type: Observational
Why Stopped: Inclusion of the last patient
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: UF 9551
Record Dates: First submitted 2016-09-02; First posted 2016-11-30 (Estimated); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Systemic Autoinflammatory Diseases (SAID)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Patients with prerequisites established jointly by the reference centers . At least 3 unexplained inflammatory access elevated CRP (C reactive protein)
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention

SUMMARY:
Main objective: To compare the efficacy of a new strategy of Next Generation Sequencing (NGS) versus a classical Sanger strategy, for the diagnosis of patients referred to the laboratory for suspected systemic autoinflammatory diseases (SAID).

Secondary objectives:

* Compare after 6 months the impact of these strategies on the establishment of an effective treatment SAID following genetic result.
* Compare the distribution of different forms of SAID found with each genetic diagnostic strategies (NGS vs classic method).

DETAILED DESCRIPTION:
Systemic autoinflammatory diseases (SAID) include a broad spectrum of pathologies of innate immunity. In recent years, numerous publications have shown the involvement of new genes in these diseases, highlighting new pathophysiological pathways (inflammasome, NFkB: nuclear factor-kappa B, interferon) and new targeted therapies (biotherapy advantageously replacing non-specific anti-inflammatory drugs). Current laboratory diagnostic strategy is based on the Sanger method, the gold standard to date, allowing the sequential analysis of some genes (usually between 1 and 4). The nonspecific nature of the clinical presentation of these diseases, the increasing number of genes involved and the low diagnostic yield obtained, make it essential to develop a new strategy, more efficient, so that the patient can benefit as soon as possible treatment suited to his pathology as soon as the gene involved is identified. The investigator had developed and validated in our genetic laboratories a new method based on the Next Generation Sequencing (NGS). A panel of 32 known or candidate SAID genes, which can be simultaneously analyzed within a time compatible with the diagnosis. The investigator wishes to highlight the benefits of this new strategy.

ELIGIBILITY:
Inclusion Criteria:

Patients with prerequisites established jointly by the reference centers:

* At least 3 unexplained inflammatory access
* Elevated C Reactive Protein
* Age of symtoms less than 30 years and validated by a physician CeréMAI (Centre de référence des maladies autoinflamatoires)

Exclusion Criteria:

* Other inflammatory disease:
* intercurrent infection
* cancer
* autoimmune disease

Ages: 3 Months to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred to the laboratory for suspected Systemic Autoinflammatory Diseases (SAID)
Sampling Method: Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2015-07-31 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Number of genetically ascertained patients using Next Generation Sequencing (NGS) vs Sanger | At time of report issue up to two years

SECONDARY OUTCOMES:
Date of introduction of relevant treatment | 6 months after report issue

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume SARRABAY, md, Principal Investigator — University Hospital, Montpellier
Locations (1):
- university Hospital Montpellier, Montpellier, France

REFERENCES:
- [Derived] Rama M, Mura T, Kone-Paut I, Boursier G, Aouinti S, Touitou I, Sarrabay G. Is gene panel sequencing more efficient than clinical-based gene sequencing to diagnose autoinflammatory diseases? A randomized study. Clin Exp Immunol. 2021 Jan;203(1):105-114. doi: 10.1111/cei.13511. Epub 2020 Sep 29. PMID 32909274